CLINICAL TRIAL: NCT04642976
Title: Prospective Evaluation of Computed Tomography Guided Ablation of Cardiac Ganglionated Plexi in Patients With Atrial Fibrillation
Brief Title: Prospective Evaluation of CT Guided Ablation of Cardiac Ganglionated Plexi
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 844182
Record Dates: First submitted 2020-11-13; First posted 2020-11-24 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Ganglionated Plexus; Cardioneural Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Atrial fibrillation ablation: All patients undergoing ablation with undergo pre-procedural CT as well as HFS mapping and ablation of GPs.
  Interventions: Device: Ganglionated Plexi mapping and ablation using Natus Cortical Stimulator and standard ablation catheters

INTERVENTIONS:
Device: Ganglionated Plexi mapping and ablation using Natus Cortical Stimulator and standard ablation catheters — Ganglionated plexi will be mapped using high frequency stimulation with standard ablation catheters attached to a Natus Cortical Stimulator for high frequency stimulation. Vagal innervation to the heart will be assessed with non-invasive Parasym tragal stimulation.
  Other Names: Vagal stimulation using Parasym tragal stimulator

SUMMARY:
Despite progress made in treating atrial fibrillation with catheter ablation, outcomes remain suboptimal with pulmonary vein isolation alone. Ablation of ganglionated plexi (GP) has been shown to be beneficial in patients with atrial fibrillation although optimal strategies of localization of these regions have yet to be determined. The investigators aim to develop a novel strategy of CT guided GP localization to guide ablation in patients with atrial fibrillation. The investigators also aim to clarify the network of innervation between GP to clarify the optimal ablation strategy. This is an observational, single-center study evaluating feasibility and efficacy of CT and high frequency stimulation (HFS) guided GP mapping and ablation in patients with AF undergoing catheter ablation with pulmonary vein isolation. Patients will undergo HFS and CT guided mapping of GPs followed by allocation into one of 8 different GP ablation approaches in a non-randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years
4. History of AF with plan to undergo catheter ablation

Exclusion Criteria:

1. Contraindication or unwillingness to undergo CT imaging or catheter ablation.
2. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with atrial fibrillation planned to undergo catheter ablation
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saman Nazarian, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atrial Fibrillation Ablation
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Atrial Fibrillation Ablation
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between HFS (High Frequency Stimulation) Response and CT Identified Epicardial Adipose Tissue.
Description: Number of patients with HFS response identified within 3 pixels (0.625x3=1.875mm) of a location where CT identified epicardial adipose tissue.
Time Frame: During Procedure
Measure: Number; unit: Number of patients with HFS response
Arm/Group | Atrial Fibrillation Ablation
Number analyzed (Participants) | 19
Number of patients with HFS response | 3

2. Secondary Outcome: HFS (High Frequency Stimulation) Response Elimination
Description: Elimination of local of HFS response following GP ablation
Time Frame: during procedure
Reporting Status: Not Posted

3. Secondary Outcome: Global Vagal Response Elimination
Description: Elimination of global vagal response to non-invasive tragal stimulation
Time Frame: This will be assessed during the procedure.
Reporting Status: Not Posted

4. Secondary Outcome: Ablation Site Changes - Amplitude of Signals
Description: Characterization of amplitude signals at sites with HFS responses and successful HFS elimination
Time Frame: This will be assessed during the procedure.
Reporting Status: Not Posted

5. Secondary Outcome: Ablation Site Changes - Duration of Signals
Description: Characterization of duration of signals at sites with HFS responses and successful HFS elimination
Time Frame: This will be assessed during the procedure.
Reporting Status: Not Posted

6. Secondary Outcome: Ablation Site Changes - Fractionation of Signals
Description: Characterization of fractionation of signals at sites with HFS responses and successful HFS elimination
Time Frame: This will be assessed during the procedure.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Atrial Fibrillation Ablation
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT04642976/Prot_SAP_000.pdf